CLINICAL TRIAL: NCT05104229
Title: SAVES-IBD: Safety & Efficacy of Aspirin vs. Standard of Care for VTE Prophylaxis After Major Surgery for Inflammatory Bowel Disease - A Pragmatic Clinical Trial
Brief Title: SAVES-IBD: Safety & Efficacy of Aspirin vs. Standard of Care for VTE Prophylaxis After IBD Surgery
Acronym: SAVES-IBD
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Limited Resources
Sponsor: Stefan Holubar MD MS FACS, FASCRS (Other)
Responsible Party: Sponsor-Investigator, Stefan Holubar MD MS FACS, FASCRS, Principal Investigator, The Cleveland Clinic
Organization: The Cleveland Clinic (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0
Record Dates: First submitted 2021-10-21; First posted 2021-11-02 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Crohn Disease; Ulcerative Colitis; Venous Thromboembolism
Keywords: surgery; prophylaxis
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Venous Thromboembolism | interventions — Aspirin; Standard of Care

STUDY DESIGN:
Intervention Model Description: Two-armed open-labeled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): standard VTE chemoprophylaxis
  Interventions: Drug: Standard of Care
- Aspirin (Experimental): Aspirin VTE chemoprophylaxis
  Interventions: Drug: Aspirin 81Mg Ec Tab

INTERVENTIONS:
Drug: Aspirin 81Mg Ec Tab — Aspirin 81Mg Ec Tab by mouth twice daily starting the day after surgery until hospital discharge, then for 30 days
  Arms: Aspirin
Drug: Standard of Care — Standard of Care VTE prophylaxis
  Arms: Standard of Care

SUMMARY:
Aim to determine if aspirin 81 mg orally twice daily is effective and safe as an extended VTE chemoprophylaxis agent after major abdominal surgery for IBD patients. Study will perform an open label trial of aspirin for VTE prophylaxis compared standard of care.

DETAILED DESCRIPTION:
Patients with inflammatory bowel disease who undergo abdominopelvic intestinal surgery are at increased risk for developing venous thromboembolism, in the form of deep vein thrombosis, pulmonary embolism and mesenteric vein thrombosis for 90-days after surgery. Despite being high-risk, the standard of care is to provide mechanical and chemoprophylaxis (unfractionated heparin or low molecular weight heparin) only while they are hospitalized. There exists randomized data, in patients who have had surgery for abdominopelvic cancer, confirming the efficacy of extended post-discharge chemoprophylaxis with either unfractionated heparin or low molecular weight heparin for 28 days after surgery, but no such data exists for IBD. There has been a resistance to adopting this for IBD patients due to compliance and cost of the daily injections. However, recently, a large, multicenter, randomized trial in >3000 patients who underwent total hip or total knee replacement found that extended aspirin (81 mg) twice daily post-discharge was both equivalent and non-inferior to prophylaxis using full-strength anticoagulation with a factor Xa inhibitor. This is a prospective, multicenter, open label clinical trial to assess the safety and efficacy of post-operative venous thromboembolism (VTE) prophylaxis with aspirin 81 mg orally twice daily for 30-days after surgery for IBD compared with controls receiving standard of care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18yrs
* Major abdominopelvic surgery with colon or rectal resection
* Preoperative diagnosis of Crohn's disease, ulcerative colitis, indeterminate colitis
* Elective surgery
* candidate for standard of care VTE prophylaxis

Exclusion Criteria:

* age < 100 yrs
* aspirin allergy
* loop ileostomy closure
* emergency surgery
* peptic ulcer disease
* cirrhosis
* bleeding or clotting disorder
* thrombocytopenia
* chronic renal insufficiency or failure
* severe anemia < 7 preoperatively
* need for therapeutic anticoagulation or anti-platelet agents post-operatively including aspirin, warfarin, heparin, clopidogrel, rivaroxaban, others

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
VTE Rate | 30-days after discharge from hospital following IBD surgery

SECONDARY OUTCOMES:
Composite of bleeding requiring transfusion or intervention | 30-days after discharge from hospital following IBD Surgery

CONTACTS AND LOCATIONS:
Overall Officials: Stefan D Holubar, MD, MS, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic Main Campus, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No